CLINICAL TRIAL: NCT05175625
Title: A Randomized, Two-Armed, Placebo-Controlled, Double-Blind, Parallel-Group Clinical Trial to Evaluate the Immunogenicity and Safety of a Booster Dose of an Adjuvanted Recombinant Spike Protein COVID-19 Vaccine (SpikoGen)
Brief Title: Immunogenicity and Safety of a Booster Dose of the SpikoGen COVID-19 Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cinnagen (Industry)
Collaborators: Vaxine Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAC.CIN.PT.BOOSTER; IRCT20150303021315N26 (Registry Identifier: Iranian Registry of Clinical Trials)
Record Dates: First submitted 2022-01-03; First posted 2022-01-04 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; Recombinant protein; Spike; Advax-SM; Advax; Vaccine; Adjuvant
MeSH Terms: conditions — COVID-19 | interventions — SARS-CoV-2 recombinant spike protein with delta inulin and CpG-ODN adjuvant vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SpikoGen COVID-19 Vaccine (Experimental)
  Interventions: Biological: SARS-CoV-2 recombinant spike protein + Advax-SM adjuvant
- Saline Placebo (Placebo Comparator)
  Interventions: Biological: Saline placebo

INTERVENTIONS:
Biological: SARS-CoV-2 recombinant spike protein + Advax-SM adjuvant — SARS-CoV-2 recombinant spike protein (25 µg) with Advax-SM adjuvant (15 mg); a single intramuscular injection into the deltoid muscle of the non-dominant arm
  Other Names: COVAX-19
  Arms: SpikoGen COVID-19 Vaccine
Biological: Saline placebo — 0.9% sodium chloride (1 mL); a single intramuscular injection into the deltoid muscle of the non-dominant arm
  Arms: Saline Placebo

SUMMARY:
This was a randomized, two-armed, double-blind, placebo-controlled trial designed to evaluate the safety and immunogenicity of a booster dose of an adjuvanted recombinant SARS-CoV-2 spike protein subunit vaccine (SpikoGen) produced by CinnaGen Co. A total of 300 adult individuals received a single dose of either the SpikoGen vaccine or the saline placebo in a 5:1 ratio at 4 to 9 months after the second dose of a COVID-19 vaccine of any type. The injection was given in the deltoid muscle of the non-dominant arm. On day 14, the trial was unblinded, and the participants in the placebo group received a booster dose of the SpikoGen vaccine. For immunogenicity assessments, blood samples were collected on days 0 and 14 from all participants and on days 90 and 180 from those in the vaccine group only. For safety assessments, all participants were followed up for six months.

Study hypotheses included:

1. A booster dose of the SpikoGen COVID-19 vaccine is safe and tolerable in adult subjects.
2. A booster dose of the SpikoGen COVID-19 vaccine induces strong immunogenicity against SARS-CoV-2 in adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years
* Willing and able to comply with all study requirements, including scheduled visits, interventions, and laboratory tests
* Healthy adults or adults in a stable medical condition, defined as not being hospitalized within 3 months prior to the screening visit
* Subjects who have received two doses of a COVID-19 vaccine of any type between 4 to 9 months before the screening visit

Exclusion Criteria:

* Subjects with signs of active SARS-CoV-2 infection at the screening visit or within 72 hours prior to the screening visit
* Subjects who have been diagnosed with a breakthrough infection after receiving two doses of a COVID-19 vaccine
* Subjects with epilepsy or a history of febrile seizures
* Subjects who receive immunosuppressive or cytotoxic medications.
* Subjects who have a history of severe allergic reactions (e.g., anaphylaxis) to the study vaccine, any components of the study interventions, or any pharmaceutical products.
* Subjects who have received any other investigational products within 30 days prior to the screening visit or intend to participate in any other clinical studies during the period of this study.
* Subjects who have received any vaccines within 28 days prior to the screening visit or intend to receive any vaccines up to day 14 of the study.
* Subjects who have any known bleeding disorders or, in the investigator's opinion, have any contraindications for an intramuscular injection.
* Female Subjects who are pregnant or breastfeeding or have planned to become pregnant within one month after the study injection.
* Subjects who have received any blood, plasma, or immunoglobulin products from 90 days prior to the screening visit or intend to receive during the study period.
* Subjects with any condition that may increase the risk of participating in the study or may interfere with the evaluation of the primary endpoints of the study in the investigator's opinion.
* Subjects who have donated ≥450 mL of blood or blood products within 28 days prior to the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with seroconversion for SARS-CoV-2 neutralizing antibodies | 14 days after the booster dose
  As measured by ELISA

SECONDARY OUTCOMES:
Incidence of solicited adverse events | For 7 days after the booster dose
  Injection site pain, erythema, swelling, and induration, axillary swelling or tenderness ipsilateral to the side of injection, fever (oral temperature), headache, fatigue, myalgia, arthralgia, nausea, vomiting, and chills, as reported by the study participants on electronic diaries, and as defined using system organ classes and preferred terms of the Medical Dictionary for Regulatory Activities (MedDRA)
Incidence of unsolicited adverse events | For 14 days after the booster dose
  As reported by the study participants on electronic diaries, and as defined using system organ classes and preferred terms of the Medical Dictionary for Regulatory Activities (MedDRA)
Incidence of serious adverse events (SAEs) and suspected unexpected serious adverse reaction (SUSARs) | For 6 months after the booster dose
  As defined using system organ classes and preferred terms of the Medical Dictionary for Regulatory Activities (MedDRA)
Geometric mean concentration (GMC) for S1 binding IgG antibodies | Days 0, 14, 90, and 180
  As measured by ELISA
Geometric mean fold rise (GMFR) for S1 binding IgG antibodies | 14 days after the booster dose
  As measured by ELISA
Percentage of participants with seroconversion for S1 binding IgG antibodies | 14 days after the booster dose
  As measured by ELISA
Percentage of participants with seroconversion for receptor-binding domain (RBD) binding IgG antibodies | 14 days after the booster dose
  As measured by ELISA
Geometric mean concentration (GMC) for receptor-binding domain (RBD) binding IgG antibodies | Days 0, 14, 90, and 180
  As measured by ELISA
Geometric mean fold rise (GMFR) for receptor-binding domain (RBD) binding IgG antibodies | 14 days after the booster dose
  As measured by ELISA
Geometric mean concentration (GMC) for SARS-CoV-2 neutralizing antibodies | Days 0, 14, 90, and 180
  As measured by ELISA
Geometric mean fold rise (GMFR) for SARS-CoV-2 neutralizing antibodies | 14 days after the booster dose
  As measured by ELISA
Change in T-cell IFN-γ secretion from baseline to 14 days after the booster dose | Days 0 and 14
  As measured by IGRA

CONTACTS AND LOCATIONS:
Overall Officials: Payam Tabarsi, M.D., Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- Orchid Life Department, Orchid Pharmed Company, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tabarsi P, Anjidani N, Shahpari R, Roshanzamir K, Fallah N, Andre G, Petrovsky N, Barati S. Immunogenicity and safety of SpikoGen(R), an adjuvanted recombinant SARS-CoV-2 spike protein vaccine as a homologous and heterologous booster vaccination: A randomized placebo-controlled trial. Immunology. 2022 Nov;167(3):340-353. doi: 10.1111/imm.13540. Epub 2022 Jul 13. PMID 35758850